CLINICAL TRIAL: NCT04385277
Title: A Pilot Study of Dinutuximab, Sargramostim (GM-CSF), and Isotretinoin in Combination With Irinotecan and Temozolomide in the Post-Consolidation Setting for High-Risk Neuroblastoma
Brief Title: Treatment With Dinutuximab, Sargramostim (GM-CSF), and Isotretinoin in Combination With Irinotecan and Temozolomide After Intensive Therapy for People With High-Risk Neuroblastoma (NBL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANBL19P1; NCI-2020-02950 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL19P1 (Other: Children's Oncology Group); ANBL19P1 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Ganglioneuroblastoma, Nodular; Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma | interventions — Specimen Handling; Biopsy; dinutuximab; 3-Iodobenzylguanidine; Irinotecan; Isotretinoin; Magnetic Resonance Spectroscopy; sargramostim; Colony-Stimulating Factors; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (temozolomide, irinotecan, dinutuximab) (Experimental): Patients receive temozolomide PO or via enteral tube daily and irinotecan IV over 90 minutes daily on days 1-5, dinutuximab IV over 10-20 hours daily on days 2-5, sargramostim SC or IV over 2 hours daily on days 6-12, and isotretinoin PO BID on days 8-21. Patients undergo MUGA during screening. Patients also undergo MRI, or CT, I23I-MIBG, or FDG-PET, BM aspiration, and BM biopsy on study. Treatment repeats every 28 days for up to 5 cycles (up to 6 cycles for isotretinoin only) in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Dinutuximab; Procedure: FDG-Positron Emission Tomography; Radiation: Iobenguane I-123; Drug: Irinotecan; Drug: Isotretinoin; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Sargramostim; Drug: Temozolomide

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo BM aspiration
Procedure: Bone Marrow Biopsy — Undergo BM biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Radiation: Iobenguane I-123 — Undergo 123I-MIBG
  Other Names: AdreView; iobenguane I 123
Drug: Irinotecan — Given IV
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Sargramostim — Given SC or IV
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Drug: Temozolomide — Given PO or via enteral tube
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial studies if dinutuximab, GM-CSF, isotretinoin in combination with irinotecan, and temozolomide (chemo-immunotherapy) can be given safely to patients with high-risk neuroblastoma after Consolidation therapy (which usually consists of two autologous stem cell transplants and radiation) who have not experienced worsening or recurrence of their disease. Dinutuximab represents a kind of cancer therapy called immunotherapy. Unlike chemotherapy and radiation, dinutuximab targets the cancer cells without destroying nearby healthy cells. Sargramostim helps the body produce normal infection-fighting white blood cells. Isotretinoin helps the neuroblastoma cells become more mature. These 3 drugs (standard immunotherapy) are already given to patients with high-risk neuroblastoma after Consolidation because they have been proven to be beneficial in this setting. Chemotherapy drugs, such as irinotecan and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. They may also affect how well immunotherapy works on neuroblastoma cells. Giving chemo-immunotherapy after intensive therapy may work better in treating patients with high-risk neuroblastoma compared to standard immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of administering dinutuximab, GM-CSF, and isotretinoin in combination with irinotecan and temozolomide in the frontline Post-Consolidation setting in patients with high-risk neuroblastoma who have undergone Induction and Consolidation therapy with tandem high-dose chemotherapy with stem cell rescue (ASCT).

SECONDARY OBJECTIVES:

I. To describe the toxicity profile of dinutuximab, GM-CSF, and isotretinoin in combination with irinotecan and temozolomide in the Post-Consolidation setting.

II. To describe the event-free survival and overall survival of patients who receive dinutuximab in combination with irinotecan and temozolomide, GM-CSF, and isotretinoin in the Post-Consolidation setting.

EXPLORATORY OBJECTIVES:

I. To describe the toxicity profiles associated with chemo-immunotherapy in the Post-Consolidation setting according to the type of prior therapy.

II. To describe response to chemo-immunotherapy in the Post-Consolidation setting using the revised International Neuroblastoma Risk Classification (INRC) in patients with evaluable or measurable disease at study entry.

III. To characterize immune and cytokine profiles in patients receiving Post-Consolidation chemo-immunotherapy.

IV. To bank serial blood samples to investigate the relationship between factors related to the tumor, host, and immune environment and clinical outcomes in patients treated with chemo-immunotherapy.

OUTLINE:

Patients receive temozolomide orally (PO) or via enteral tube daily and irinotecan intravenously (IV) over 90 minutes daily on days 1-5, dinutuximab IV over 10-20 hours daily on days 2-5, sargramostim subcutaneously (SC) or IV over 2 hours daily on days 6-12, and isotretinoin PO twice daily (BID) on days 8-21. Patients undergo multigated acquisition scan (MUGA) during screening. Patients also undergo magnetic resonance imaging (MRI), or computed tomography (CT), iobenguane I-123 (123I-MIBG), or fludeoxyglucose F-18-positron emission tomography (FDG-PET), bone marrow (BM) aspiration, and BM biopsy on study. Treatment repeats every 28 days for up to 5 cycles (up to 6 cycles for isotretinoin only) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be < 31 years of age at the time of enrollment.
* Patients must have a diagnosis of neuroblastoma or ganglioneuroblastoma (nodular) (verified by tumor pathology analysis or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites at the time of diagnosis) and have been designated as having high-risk disease based on Children's Oncology Group (COG) risk classification. The following disease groups are eligible:

  * Patients with International Neuroblastoma Risk Group (INRG) Stage M disease with any of the following features:

    * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of additional biologic features; OR
    * Age > 547 days at the time of diagnosis regardless of biologic features; OR
    * Age 365-547 days at the time of diagnosis with tumors with unfavorable histology and/or deoxyribonucleic acid (DNA) index = 1
  * Patients with INRG Stage MS disease with MYCN amplification
  * Patients with INRG Stage L2 disease with either of the following features:

    * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of additional biologic features; OR
    * Age > 547 days at the time of diagnosis with MYCN non-amplified tumors with unfavorable histology
  * Note: Patients observed or patients treated with a single cycle of chemotherapy per a low or intermediate risk neuroblastoma regimen (e.g., as per ANBL0531, ANBL1232 or similar) for what initially appeared to be non-high-risk disease but subsequently found to meet criteria will also be eligible
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years
* Prior therapy

  * All patients must have completed high-risk Induction therapy with 4-6 cycles of chemotherapy
  * After completion of Induction therapy, patients may have received no more than 4 cycles of bridging chemotherapy or chemo-immunotherapy prior to ASCT
  * Patients cannot have previously progressed on immunotherapy with dinutuximab or other anti-GD2 monoclonal antibody
  * All patients must have had undergone surgical resection of their primary tumor as part of frontline therapy. Exceptions to this requirement include patients who had a complete response to Induction chemotherapy, patients with no identifiable primary tumor, and patients for whom the institutional surgical team determined that potential risks outweighed potential benefits of resection
  * All patients must have undergone tandem high-dose chemotherapy with ASCT as part of Consolidation
  * Patients must enroll between day +56 and day +200 from the peripheral blood stem cell (PBSC) infusion following the last dose of high-dose chemotherapy during Consolidation
  * All patients must have undergone external beam radiation therapy. Exceptions to this requirement include patients who had no identifiable primary tumor and no persistent metastatic disease at the end of Induction. For patients who received radiotherapy, at least 7 days must have elapsed between completion of radiotherapy and enrollment on this study
* Patients must not have received long-acting myeloid growth factors (e.g., Neulasta) within 14 days of entry on this study. Seven days must have elapsed since administration of a short-acting myeloid growth factor
* Peripheral absolute neutrophil count (ANC) >= 750/uL
* Platelet count >= 50,000/uL (transfusion independent for >= 7 days)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2, or a serum creatinine based on age/gender as follows:

  * Age: Maximum Serum Creatinine (mg/dL)
  * 6 months to < 1 year: 0.5 (male and female)
  * 1 to < 2 years: 0.6 (male and female)
  * 2 to < 6 years: 0.8 (male and female)
  * 6 to < 10 years: 1 (male and female)
  * 10 to < 13 years: 1.2 (male and female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)

    * Note: Patients with history of transplant associated-thrombotic microangiopathy (TA-TMA) must have a creatinine clearance or radioisotope GFR at baseline to assess renal function and must meet the above criteria
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5.0 x ULN for age (=< 225 U/L)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by echocardiogram or radionuclide angiogram
* Absence of dyspnea at rest
* If pulmonary function tests (PFTs) are performed, forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) must be > 60%
* No clinical evidence of active central nervous system (CNS) disease at the time of study enrollment
* Patients with seizure disorder may be enrolled if on non-enzyme-inducing anticonvulsants and well controlled
* CNS toxicity from prior therapy =< grade 2

Exclusion Criteria:

* Patients must not have had progressive disease (PD) per the revised International Neuroblastoma Risk Criteria (INRC) since the initial diagnosis of high-risk neuroblastoma

  * Exception: Progressive disease within the first 2 cycles of Induction chemotherapy consisting of cyclophosphamide and topotecan is allowed. Patients with progression subsequent to initial cyclophosphamide and topotecan cycles are excluded
* Patients may not have received additional systemic cancer-directed therapy following completion of the last planned high-dose chemotherapy with ASCT prior to enrollment on this trial
* Patients may not have received iodine-131 (131I)-metaiodobenzylguanidine (MIBG) therapy at any time prior to enrollment on this trial
* Patients who received single (rather than tandem) high-dose chemotherapy with ASCT are excluded
* Patients cannot be receiving other ongoing anticancer therapy
* Patients who were enrolled onto ANBL1531 AND underwent arm assignment are not eligible. Patients who enrolled onto ANBL1531 who declined second consent may be eligible for ANBL19P1 if all other criteria are met
* Patients enrolled onto ANBL17P1 are not eligible
* Patients must have been off pharmacologic doses of systemic steroids for at least 7 days prior to enrollment
* Patients who require or are likely to require pharmacologic doses of systemic corticosteroids while receiving treatment on this study are ineligible. The only exception is for patients known to require 2 mg/kg or less of hydrocortisone (or an equivalent dose of an alternative corticosteroid) as premedication for blood product administration in order to avoid allergic transfusion reactions

  * Note: The use of conventional doses of inhaled steroids for the treatment of asthma is permitted, as is the use of physiologic doses of steroids for patients with known adrenal insufficiency
* Patients on any other immunosuppressive medications (e.g., cyclosporine, tacrolimus) are not eligible. However, prior or planned concomitant treatment with eculizumab is permitted (e.g., treatment of TA-TMA)
* Patients must not have received enzyme-inducing anticonvulsants including phenytoin, phenobarbital, valproic acid, or carbamazepine for at least 7 days prior to study enrollment

  * Note: Patients receiving non-enzyme inducing anticonvulsants such as gabapentin or levetiracetam are eligible
* Patients must not have received drugs that are strong inducers or inhibitors of CYP3A4 within 7 days prior to study enrollment
* Patients must not have been diagnosed with myelodysplastic syndrome or with any malignancy other than neuroblastoma
* Patients with symptoms of congestive heart failure are not eligible
* Patients with moderate or large pericardial effusions are not eligible
* Patients must not have >= grade 2 diarrhea
* Patients must not have uncontrolled infection
* Patients with a history of grade 4 allergic reactions to anti-GD2 antibodies or reactions that required discontinuation of the anti-GD2 therapy are not eligible
* Patients with a significant intercurrent illness (any ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and that is expected to interfere with the action of study agents or to significantly increase the severity of the toxicities experienced from study treatment are not eligible
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2027-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ami V Desai, Principal Investigator — Children's Oncology Group
Locations (77):
- United States (70):
  - Banner Children's at Desert, Mesa, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - NYU Winthrop Hospital, Mineola, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- IWK Health Centre, Halifax, Nova Scotia, Canada
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with newly diagnosed high-risk Neuroblastoma enrolled between 12/31/2020 and 6/27/2022 across 22 institutions.
Groups:
- Treatment (Temozolomide, Irinotecan, Dinutuximab): Patients receive temozolomide PO or via enteral tube daily and irinotecan IV over 90 minutes daily on days 1-5, dinutuximab IV over 10-20 hours daily on days 2-5, sargramostim SC or IV over 2 hours daily on days 6-12, and isotretinoin PO BID on days 8-21. Patients undergo MUGA during screening. Treatment repeats every 28 days for up to 5 cycles (up to 6 cycles for isotretinoin only) in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI, or CT, I23I-MIBG, or FDG-PET, BM aspiration, and BM biopsy on study.
Period: Overall Study
Arm/Group | Treatment (Temozolomide, Irinotecan, Dinutuximab)
Started | 41
Completed | 36
Not Completed | 5
Not completed — Physician Decision | 2
Not completed — Ineligible | 1
Not completed — Patient/Parent Refusal | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Temozolomide, Irinotecan, Dinutuximab)
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.74 (2.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 26
  More than one race | 1
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 34
  New Zealand | 4
  Australia | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Complete 5 Cycles of Dinutuximab + Chemotherapy Without Progressive Disease (PD)
Description: Will be assessed by estimation of the feasibility therapy completion rate together with a 95% Wilson confidence interval (CI).
Time Frame: Within 30 weeks from the date of first treatment
Population: All eligible patients who receive at least one dose of dinutuximab in combination with irinotecan and temozolomide, GM-CSF, and isotretinoin
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Temozolomide, Irinotecan, Dinutuximab)
Number analyzed (Participants) | 40
Percentage of patients | 87.50 [73.89 to 94.54]

2. Secondary Outcome: Event-free Survival (EFS)
Description: EFS Kaplan-Meier estimates will be generated.
Time Frame: From the time of start of protocol therapy to the occurrence of disease relapse or progression, secondary malignancy, or death, assessed at 1 year.
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Temozolomide, Irinotecan, Dinutuximab)
Number analyzed (Participants) | 40
percentage of participants | 90.0 [80.71 to 99.29]

3. Secondary Outcome: Overall Survival (OS)
Description: OS Kaplan-Meier estimates will be generated.
Time Frame: From the time of start of protocol therapy to death, assessed at 1 year.
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Temozolomide, Irinotecan, Dinutuximab)
Number analyzed (Participants) | 40
percentage of participants | 97.5 [92.66 to 100]

ADVERSE EVENTS:
Time Frame: Enrollment up to 2 years after finishing protocol therapy
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Temozolomide, Irinotecan, Dinutuximab)
All-Cause Mortality (participants affected / at risk) | 2/40
Serious Adverse Events (participants affected / at risk) | 3/40
Other Adverse Events (participants affected / at risk) | 34/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temozolomide, Irinotecan, Dinutuximab) (N=40)
Death NOS (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Temozolomide, Irinotecan, Dinutuximab) (N=40)
Anemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Gastrointestinal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fever (General disorders) | 17
Pain (General disorders) | 12
Anaphylaxis (Immune system disorders) | 1
Enterocolitis infectious (Infections and infestations) | 4
Infections and infestations - Other, specify (Infections and infestations) | 4
Otitis media (Infections and infestations) | 1
Sepsis (Infections and infestations) | 7
Upper respiratory infection (Infections and infestations) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 4
GGT increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 12
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 12
Platelet count decreased (Investigations) | 8
White blood cell decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 15
Iron overload (Metabolism and nutrition disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Seizure (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT04385277/Prot_SAP_000.pdf